CLINICAL TRIAL: NCT04649489
Title: A Multicenter, Randomized, Open-label Study Evaluating the Efficacy and Safety of Hepatic Resection for Hepatocellular Carcinoma With Venous Thrombosis After Initial Atezolizumab Plus Bevacizumab Treatment
Brief Title: A Study to Evaluate Efficacy and Safety of Hepatic Resection for Liver Cancer With PVTT, HVTT or IVCTT After Initial Ate/Bev
Acronym: TALENTOP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jia Fan (Other)
Responsible Party: Sponsor-Investigator, Jia Fan, Doctor of hospital, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML42435
Record Dates: First submitted 2020-11-12; First posted 2020-12-02 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (experimental arm) (Experimental): hepatic resection with post-operative atezolizumab 1200mg and bevacizumab 15mg/kg, both administered by IV infusion on Day 1 of each 21-day cycle
  Interventions: Procedure: Surgery followed by atezolizumab and bevacizumab
- Arm B (control arm) (Active Comparator): atezolizumab 1200mg and bevacizumab 15mg/kg, both administered by IV infusion on Day 1 of each 21-day cycle
  Interventions: Drug: Atezolizumab & Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab & Bevacizumab — atezolizumab 1200mg and bevacizumab 15mg/kg
  Other Names: Bevacizumab
  Arms: Arm B (control arm)
Procedure: Surgery followed by atezolizumab and bevacizumab — hepatic resection with post-operative atezolizumab 1200mg and bevacizumab 15mg/kg
  Other Names: Atezolizumab; Bevacizumab
  Arms: Arm A (experimental arm)

SUMMARY:
The treatment strategies for HCC with PVTT is still controversial, and differ substantially between the west and the east. According to western guidelines, including those of the EASL, BCLC, and AASLD, PVTT is regarded as a contra-indication to initial surgery or transarterial chemoembolization.

At present, there is still no consensus on the diagnosis and treatment standards of HCC with HVTT/IVCTT. European and American guidelines for liver cancer use The Barcelona Clinic Liver Cancer (BCLC) staging as the standard and classify liver cancer with HVTT/IVCTT into the advanced stage. Molecular targeted drugs such as sorafenib and lenvatinib are recommended to the patients in this phase as first-line treatment drugs and methods. In this regard, experts in China and Southeast Asian countries still have different opinions. They believe that surgery, transarterial chemoembolization (TACE), radiotherapy, and combined treatment with multiple treatment methods can achieve more satisfactory results.

HCC with VTT consists of heterogeneous populations with different disease behaviors and prognoses. As a result of recent concept evolution and advances in surgical techniques and perioperative management, emerging evidence shows that selected patients with PVTT may benefit from more aggressive treatment modalities, which are recommended for by Chinese, Japanese, South Korean, and Asia Pacific clinical practice guidelines. A national survey from Japan showed median overall survival with liver resection treatment to be 1.77 years longer than with nonresection therapies, which included TACE, radiotherapy, sorafenib, or conservative treatment (2.87 years vs 1.10 years, respectively; p<0.001). After propensity-score matching of patient baseline characteristics, median overall survival since diagnosis in the liver resection group was 0.88 years longer than in the non-resection group. In a large-scale, multicentre, propensity-score matched analysis from China, surgery was the best treatment for patients with Cheng's type I and II PVTT with Child-Pugh A and selected B liver function. Median overall survival after liver resection (745 of 1580 patients) was 15.9 months (95% CI 13.3-18.5 months) for Cheng's type I PVTT and 12.5 months (10.7-14.3 months) for Cheng's type II PVTT. Thus, aggressive surgical resection in selected patients with HCC with vascular invasion, as proposed by several tertiary health-care centers in the east, seems to be reasonable.

Currently, there are no dedicated clinical trials to study the value of hepatic resection in this population. Furthermore, cumulative evidence indicates that long-term overall survival after hepatic resection alone remains unsatisfactory because of the high rate of tumor recurrence and correspondingly low rate of disease-free survival. The combination of perioperative therapies may be more efficacious to improve the prognosis in selected population. More high-level evidence of novel multimodality treatment should be generated.

This trial will enroll HCC patients with PVTT CNLC Stage IIIa, who have no prior anti-cancer treatment. Given the poor prognosis and limited treatment options for these patients, this population is considered appropriate for trials of more aggressive and novel therapeutic candidates in the initial treatment setting. The benefit risk profile for hepatic resection combined with perioperative atezo/bev in this patient population is expected to be favorable.

DETAILED DESCRIPTION:
This is a multicenter, open-label, two-arm, randomized study designed to evaluate the efficacy and safety of surgical resection plus peri-operative atezo/bev compared with continuous systemic atezo/bev in HCC patients with VTT and without EHS.

Initially eligible patients will be enrolled into induction phase, during which they will receive 3 cycles of atezo/bev and 1 cycle of atezo alone as primary systemic therapy. Tumor response assessment using computed tomography (CT) and/or magnetic resonance imaging (MRI) will be conducted by the Independent-Review Facility (IRF) according to RECIST v1.1 after cycle 2 and cycle 4.

Only those patients who are assessed as partial response (PR) or stable disease (SD) and considered suitable for curative hepatic resection will be randomized in a 1:1 ratio to one of the following two arms:

* Arm A (experimental arm): hepatic resection with post-operative atezolizumab 1200mg and bevacizumab 15mg/kg, both administered by IV infusion on Day 1 of each 21-day cycle
* Arm B (control arm): atezolizumab 1200mg and bevacizumab 15mg/kg, both administered by IV infusion on Day 1 of each 21-day cycle

Randomization will be performed after the second tumor assessment and stratified according to the following stratification factors:

* Tumor response: target lesion reduction (maximum diameter reduction ≥10% compared with the entry baseline) vs non-reduction
* Eastern Cooperative Oncology Group (ECOG) performance status: 0 vs 1 Those patients who are assessed as disease progression (PD) or complete response (CR) and/or not suitable for curative hepatic resection will be excluded from randomization and treated according to local practice (Patients without PD may continue atezo/bev treatment at investigators' discretion).

In Arm A, hepatic resection surgery will be performed 0-2 weeks after the randomization. Surgical approaches will be tailored to the individual patient according to local standards with the goal of achieving R0 resection. The first administration of postoperative atezo/bev treatment is recommended to start within 4-6 weeks after surgery, requiring full recovery from the surgery prior to post-operative atezo/bev treatment, including:

* Adverse events emerged from prior treatment, if any, should have been recovered to meet the requirements of atezo/bev treatment according to investigator's judgement.
* No significant medical events (e.g., gastrointestinal [GI] bleeding, cardiac events, hepatorenal syndrome, biliary fistula, serious infection, etc.) during or after the surgery procedure Treatment with atezo/bev will continue until loss of clinical benefit (determined by the investigator), or unacceptable toxicity, withdrawal of ICF, death, or the study is terminated by the Sponsor, whichever occurs first. For Arm A, whether to continue atezo/bev treatment will be determined by the investigator at the end of the 12-month treatment period if none of the above occurs.

Tumor assessments will be performed in induction phase after cycle 2 and cycle 4 (randomization baseline), and in treatment period at regular intervals (Arm A will receive tumor assessment at the first dose of postoperative treatment (±3 days）and every 9 weeks (±7 days）thereafter. Arm B every 9 weeks (±7 days）thereafter ). Additional scans will be performed as clinically indicated. Following completion or discontinuation of the treatment, information on recurrence or disease progression, survival and subsequent anti-cancer therapies will be collected until death, loss to follow-up, withdrawal of ICF or study termination by Sponsor, whichever occurs first. In the absence of disease recurrence or progression, tumor assessments should continue regardless of whether patients start a new anti-cancer therapy, until documented treatment failure events, withdrawal of ICF or study termination. All patients will be followed for survival unless consent is withdrawn.

Patients who withdraw from the study will not be replaced. An IRF will be used to enable centralized, independent reviews of images and other clinical data (e.g., histopathology, tumor markers etc.) used for assessment of HCC response, recurrence and disease progression. IRF reviews will be performed prior to the pre-specified efficacy analyses. IRF membership and procedures will be detailed in an IRF Charter.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Aged ≥18 years at time of signing ICF
3. Ability to comply with the study protocol, in the investigator's judgment
4. Documented diagnosis of HCC confirmed by histology/cytology or clinically by AASLD criteria in cirrhotic patients - Patients without cirrhosis require histological confirmation of diagnosis.
5. No prior anti-tumor treatment (including both local-regional and systemic therapies) for HCC

   * Previous use of herbal therapies/traditional Chinese medicines (TCM) with anti-cancer activity included in the label is allowed, provided that these medications are discontinued at least 7 days prior to enrollment.
6. Presence of PVTT, determined based on the radiological findings, including Vp1 (third-order branch of portal vein) to Vp4 (main trunk/collateral branch of portal vein) according to the Japanese staging system or Presence of HVTT or IVCTT, without atrium tumor thrombosis, determined based on the radiological findings
7. Remnant liver volume-to-total liver volume (RLV%) ≥ 25%
8. At least one measurable lesion (per RECIST v1.1) untreated lesion
9. ECOG performance status of 0 or 1 within 7 days prior to study entry
10. Child-Pugh class A within 7 days prior to study entry
11. Life expectancy ≥12 weeks
12. Adequate hematologic and end-organ function, defined by the following laboratory test results, obtained within 14 days prior to initiation of induction treatment unless otherwise specified:

    - Absolute neutrophil count (ANC)≥1.5x109/L (1500/uL) without granulocyte colony stimulating factor support

    - Lymphocyte count ≥0.5x109/L (500/uL)

    - Platelet count ≥75x109/L (75,000/uL) without transfusion
    * Hemoglobin ≥90 g/L (9 g/dL). Patients may be transfused to meet this criterion.
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤5x upper limit of normal (ULN)
    * Serum total bilirubin ≤3x ULN
    * Serum albumin ≥28 g/L (2.8 g/dL)
    * Serum creatinine (SCr) ≤1.5 x ULN or Creatinine clearance (CCr) ≥ 50mL/min (calculated using the Cockcroft-Gault formula):

      (140-age) x Weight (kg) CCr (ml/min) = --------------------------------- (Female x 0.85) 72 x SCr (mg/dL) (140-age) x Weight (kg) OR CCr (ml/min) = ----------------------------------- (Female x 0.85) 0.818 x SCr (umol/L)
    * For patients not receiving therapeutic anticoagulation: international normalized ratio (INR) or activated partial prothrombin time (aPTT) ≤ 1.2 x ULN
    * Urine dipstick for proteinuria < 2+ (within 7 days prior to Day 1 of Cycle 1) Patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours.
13. Resolution of any acute, clinically significant treatment-related toxicity from prior therapy to Grade ≤ 1 prior to study entry, with the exception of alopecia
14. Negative human immunodeficiency virus (HIV) test at screening
15. Documented virology status of hepatitis, as confirmed by screening hepatitis B virus (HBV) and hepatitis C virus (HCV) serology tests
16. For patients with positive HBV DNA/HCV RNA, anti-HBV/HCV thrapies are coontinued during study (base on local care of stanstand)
17. For women of childbearing potential, agreement (by patient) to remain abstinent (refrain from heterosexual intercourse) or to use contraceptive methods as defined below:

    * Women must remain abstinent or use highly effective form(s) of contraception (i.e., one that results in a low failure rate [<1% per year] when used consistently and correctly) while they are receiving atezolizumab and bevacizumab and for at least 5 months after the final dose of atezolizumab and 6 months after the final dose of bevacizumab. Women must refrain donating eggs during this same period.
    * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgical sterilization (i.e., removal of ovaries, fallopian tubes and/or uterus), or other causes as determined by the investigator (e.g., Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
    * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
18. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

    * With female partners of childbearing potential or pregnant female partners, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of <1% per year during the treatment period and for at least 6 months after the final dose of bevacizumab to avoid exposing the embryo. Men must refrain from donating sperm during this same period
    * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of preventing drug exposure. If required per local guidelines or regulations, locally recognized acceptable methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

Patients must meet the following additional criteria for study randomization:

18. Tumor assessed as PR or SD after 4 cycles of atezo/bev treatment as determined by the IRF according to RECIST v1.1 19. Feasibility for curative hepatic resection as assessed by the investigator 20. Physical condition and organ function allowing to undergo appropriate surgical management or atezo/bev treatment according to investigator's judgement.

21. Treatment emerged adverse events during induction phase, if any, should have been recovered to meet the requirements of surgical or atezo/bev treatment according to investigator's judgement.

22. Agreement and ability to comply with the treatment of Arm A or Arm B in the investigator's judgment

Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
2. Evidence of EHS, as confirmed by CT and/or MRI scans of the chest, abdomen, and pelvis
3. Evidence of HCC disease progression or complete remission prior to randomization
4. Clinically significant ascites
5. History of hepatic encephalopathy
6. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding

   * Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of atezo/bev treatment do not need to repeat the procedure.
7. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism who are on thyroidreplacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

     * Rash must cover < 10% of body surface area.
     * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
     * There is no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the 12 months prior to Day 1 of Cycle 1.
8. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
9. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to Day 1 of Cycle 1, unstable arrhythmia, or unstable angina
10. History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
11. Active tuberculosis
12. Severe infection within 4 weeks prior to Day 1 of Cycle 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
13. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to Day 1 of Cycle 1

    * Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
14. Prior allogeneic stem cell or solid organ transplantation
15. On the waiting list for liver transplantation
16. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
17. Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the final dose of atezolizumab or within 6 months after the final dose of bevacizumab

    * Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to Day 1 of Cycle 1.
18. Co-infection with HBV and HCV

    * Patients with a history of HCV infection but who are negative for HCV RNA by polymerase chain reaction will be considered to be negative for HCV infection.
19. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium, > 12mg/dL, or corrected serum calcium > ULN)
20. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
21. Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulations
22. Any prior treatment for HCC, including systemic therapy (including investigational agents) and locoregional therapy such as TACE

    * Prior use of herbal therapies or traditional Chinese medicines with anti-cancer activity included in the label is allowed, but such therapies must be discontinued at least 7 days prior to study entry and are prohibited during the study.
23. Treatment with a live, attenuated vaccine within 4 weeks prior to Day 1 of Cycle 1, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
24. Treatment with investigational therapy within 4 weeks prior to Day 1 of Cycle 1
25. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
26. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin-2) within 4 weeks or 5 drug elimination half-lives (whichever is longer) prior to Day 1 of Cycle 1
27. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor-α [TNF-α agents) within 2 weeks prior to Day 1 of Cycle 1, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor approval has been obtained.
    * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
28. Inadequately controlled arterial hypertension (defined as systolic blood pressure [BP] > 150 mmHg and/or diastolic BP > 100 mmHg), based on an average of at least three BP readings at two or more sessions

    * Anti-hypertensive therapy to achieve these parameters is allowed.
29. History of hypertensive crisis or hypertensive encephalopathy
30. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of Cycle 1 Clinical Study
31. History of hemoptysis (> 2.5 mL of bright red blood per episode) within 1 month prior to Day 1 of Cycle 1
32. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
33. Current or recent (within 10 days of Day 1 of Cycle 1) use of aspirin (> 325 mg/day) or current or recent treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol
34. Current or recent (within 10 days prior to Day 1 of Cycle 1) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose

    * Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR and aPTT is within normal limits (according to institutional standards) within 14 days prior to Day 1 of Cycle 1.
    * Prophylactic use of low-molecular-weight heparin (LMWH) (i.e., enoxaparin 40 mg/day) is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.
35. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 3 days prior to Day 1 of Cycle 1
36. History of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intraabdominal abscess within 6 months prior to Day 1 of Cycle 1
37. Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
38. Serious, non-healing or dehiscing wound, active ulcer, or untreated bone fracture
39. Major surgical procedure within 4 weeks prior to Day 1 of Cycle 1 or anticipation of need for a major surgical procedure during the study
40. History of intra-abdominal inflammatory process within 6 months prior to Day 1 of Cycle 1, including, but not limited to, peptic ulcer disease, diverticulitis, or colitis
41. History of intestinal obstruction and/or clinical signs or symptoms of GI obstruction including sub-occlusive disease related to the underlying disease or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding prior to initiation of study treatment Patients with signs/symptoms of sub-/occlusive syndrome/intestinal obstruction at time of initial diagnosis may be enrolled if they had received definitive (surgical) treatment for symptom resolution.
42. Radiotherapy within 28 days and abdominal/ pelvic radiotherapy within 60 days prior to initiation of study treatment.
43. Chronic daily treatment with a non-steroidal anti-inflammatory drugs (NSAIDs)

    * Occasional use of NSAIDs for the symptomatic relief of medical conditions such asheadache or fever is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
TTF | 24 months
  Time-to-treatment failure (TTF) after randomization, defined as the time from randomization to the first documented treatment failure (i.e., local recurrence or progression, EHS, or death from any cause). Tumor response will be determined by the IRF according to RECIST v1.1

SECONDARY OUTCOMES:
OS | 24 months
  Overall survival (OS) after randomization, defined as the time from randomization to death from any cause
OS rate | 24 months
  OS rate at 12 months, 18 months and 24 months, defined as the proportion of patients who have not experienced death from any cause at 12, 18 and 24months after randomization, respectively
TTF | 24 months
  TTF after randomization as determined by the investigator according to RECIST v1.1
TTF | 24 months
  TTF after randomization as determined by the IRF and the investigator according to HCC mRECIST
Time to EHS | 24 months
  Time to EHS after randomization, defined as the time from randomization to first appearance of EHS, as determined by the IRF and the investigator

OTHER OUTCOMES:
AE/ADR | 24 months
  Nature, incidence, severity and seriousness of the adverse events/ADR. Adverse events are graded according to the NCI-CTCAE (Version 5.0)
RFS | 24 months
  Recurrence-free survival (RFS) after randomization (Arm A), defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC as determined by the IRF and the investigator, or death from any cause (whichever occurs first)
TTR | 24 months
  Time-to-Recurrence (TTR) after randomization (Arm A), defined as the time from randomization to the first documented occurrence of local, regional, or metastatic HCC, as determined by the IRF and the investigator
R0 rate | 24 months
  R0 rate (Arm A), defined as the proportion of patients who accomplish the complete resection of tumor with pathologically confirmed negative margin
pCR rate | 24 months
  Pathological complete regression (pCR) rate (Arm A), defined as the proportion of patients with no evidence of vital residual tumor cells on the complete resected specimen. pCR status will be analyzed by local pathologists at each site
ORR | 24 months
  Objective response rate (ORR) during atezo/bev treatment in induction phase before randomization and in Arm B after randomization, defined as the proportion of patients with a complete response (CR) or partial response (PR), as determined by the IRF and the investigator according to RECIST v1.1 and HCC mRECIST

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Fudan University
Locations (23):
- China (23):
  - Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality
  - Beijing Cancer Hospital, Beijing
  - Cancer Hospital Chinese Academy of Medical Science, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking Univerty People's Hospital, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Provincial Hospital, Fuzhou
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - The Second Affiliated Hospital Kunming Medical University, Kunming
  - The First Hospital of Lanzhou University, Lanzhou
  - Jiangsu Provine People Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - The First Affiliated Hospital Of Guangxi Medical University, Nanning
  - Shanghai Jiao Tong University Ruijin Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Tongji Hospital of Tongji Medical College of HUST, Wuhan
  - Henan Province People Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: Undecided